CLINICAL TRIAL: NCT01792700
Title: Long-term Follow up Helicobacter Pylori Reinfection Rate After Second-Line Treatment: Bismuth-Containing Quadruple Therapy Versus Moxifloxacin-Based Triple Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Nayoung Kim, Department of Internal Medicine, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-0603/031-013
Record Dates: First submitted 2013-02-12; First posted 2013-02-15 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Helicobacter Infections
MeSH Terms: conditions — Helicobacter Infections | interventions — Esomeprazole; Metronidazole; Tetracycline; Moxifloxacin; Amoxicillin

ARMS (2):
- MEA (Active Comparator): MEA: moxifloxacin (400 mg q.d.), esomeprazole (20 mg b.i.d), and amoxicillin (1000 mg b.i.d.)
  Interventions: Drug: esomeprazole; Drug: moxifloxacin; Drug: amoxicillin
- EBMT (Active Comparator): EBMT: esomeprazole (20 mg b.i.d), tripotassium dicitrate bismuthate (300 mg q.i.d), metronidazole (500 mg t.i.d), and tetracycline (500 mg q.i.d)
  Interventions: Drug: esomeprazole; Drug: tripotassium dicitrate bismuthate; Drug: metronidazole; Drug: tetracycline

INTERVENTIONS:
Drug: esomeprazole
Drug: tripotassium dicitrate bismuthate
  Arms: EBMT
Drug: metronidazole
  Arms: EBMT
Drug: tetracycline
  Arms: EBMT
Drug: moxifloxacin
  Arms: MEA
Drug: amoxicillin
  Arms: MEA

SUMMARY:
patients who had failed previous H. pylori eradication on standard triple therapy were randomized into two regimens: 1, esomeprazole (20 mg b.i.d), tripotassium dicitrate bismuthate (300 mg q.i.d), metronidazole (500 mg t.i.d), and tetracycline (500 mg q.i.d) (EBMT) or 2, moxifloxacin (400 mg q.d.), esomeprazole (20 mg b.i.d), and amoxicillin (1000 mg b.i.d.) (MEA). At four weeks after completion of eradication therapy, H. pylori tests were performed with 13C urea breath test (UBT) or invasive tests (Giemsa histology, CLO test, and culture). In patients who maintained continuous H. pylori negativity for the first year after eradication therapy, H. pylori status was assessed every year. For the evaluation of risk factors of reinfection, gender, age, clinical diagnosis, histological atrophic gastritis or intestinal metaplasia were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients were considered persistent H. pylori infection if 13C-urea breath test (UBT) or invasive H. pylori test (Giemsa histology, CLO test, culture) were positive despite PPI-based triple therapy.

Exclusion Criteria:

* Patients were excluded from the study if they had a history of renal or hepatic impairment, previous gastric surgery, pregnancy or lactation, therapy with steroids or non-steroidal anti-inflammatory drugs, or therapy with a proton pump inhibitor (PPI) or antibiotics within four weeks of entry.

Ages: 23 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 648 (Actual)
Dates: Start 2003-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Helicobacter pylori reinfection rate | From date of randomization until the date of first documented reinfection of Helicobacter pylori, whichever came first, assessed up to 90 months

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Kim MS, Kim N, Kim SE, Jo HJ, Shin CM, Park YS, Lee DH. Long-term follow up Helicobacter Pylori reinfection rate after second-line treatment: bismuth-containing quadruple therapy versus moxifloxacin-based triple therapy. BMC Gastroenterol. 2013 Sep 19;13:138. doi: 10.1186/1471-230X-13-138. PMID 24050512